CLINICAL TRIAL: NCT01742754
Title: Evaluation of Durability of Fecal Microbiota Transplantation in Patients With Mild to Moderate Ulcerative Colitis
Brief Title: Fecal Microbiota Transplantation for Ulcerative Colitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: IND required by the FDA for all future FMTs.
Sponsor: University of Washington (Other)
Collaborators: The Broad Foundation (Other)
Responsible Party: Principal Investigator, Timothy Zisman, Assistant Professor of Medicine, Medicine/Division of Gastroenterology, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 41454-K
Record Dates: First submitted 2012-11-29; First posted 2012-12-05 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fecal Microbiota Transplantation (Experimental): Fecal Microbiota Transplantation by colonoscopic delivery of stool to the right colon.
  Interventions: Other: Fecal Microbiota Transplantation

INTERVENTIONS:
Other: Fecal Microbiota Transplantation — Fecal microbiota transplantation by colonoscopic administration of 300cc of fecal slurry from healthy donor to the right colon.

SUMMARY:
Fecal microbiota therapy (FMT) is an emerging treatment for gastrointestinal disorders marked by an imbalance in the intestinal microbial flora (dysbiosis). It is hypothesized to work by shifting the recipient's microbiota toward a eubiotic microbial community that resists colonization by pathogenic organisms or decreases its inherent inflammatory properties. Several studies now report its efficacy in treatment of severe Clostridium difficile colitis. Preliminary studies using FMT in Ulcerative Colitis (UC) have also met with some success. This is corroborated by several lines of evidence suggesting dysbiosis plays an important role in UC pathogenesis. While a recent study using FMT in patients with irritable bowel syndrome (IBS) and constipation found transplants persist for up to 2 years, the extent to which the microbiota is alterable in UC is not known. Indeed, there may be particular genetic or immunologic factors in UC leading to selection pressure preventing a change in the microbiota. As an initial step into investigating the potential efficacy of stool transplants for Ulcerative Colitis (UC), the investigators propose to determine the feasibility and stability of transplanted microbiota in a series of 10 patients with mild to moderate UC.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate UC.

Exclusion Criteria:

* Antibiotic exposure in the last 3 months.
* Biologic or immunomodulatory therapy within the last 3 months.
* Corticosteroid therapy or probiotics within the last 2 weeks.
* Severely active disease (defined as Mayo scores of 10 or greater, or patients with endoscopic disease activity scores of 3 or greater).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-10; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Successful engraftment of donor fecal microbiota at 4 weeks post-transplantation. | 4 weeks
  Metagenomic shotgun sequencing using Iluminia technology will be used to evaluate for engraftment. Metagenomic data will be analyzed using CompareReads. A % similarity to the recipient > than % similarity to the donor will be defined as engraftment.

SECONDARY OUTCOMES:
Engraftment of fecal microbiota transplantation at 7 days. | 7 days
  As in primary aim but at 7 days.
Durability of Fecal Microbiota Transplantation at 12 weeks | 12 weeks
  As in primary aim but at 12 weeks.
Clinical remission at 4 weeks. | 4 weeks
  Defined as Mayo score <=2 with no subscore >1
Clinical remission at 12 weeks. | 12 weeks
  Defined as Mayo score <=2 with no subscore >1
Endoscopic remission at 4 weeks. | 4 weeks
  Mayo endoscopy scope of 0.
Number of patients with worsened disease. | 4 weeks.
  Increase in Mayo score of >2.
Number of adverse events. | 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy L Zisman, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Background] Damman CJ, Miller SI, Surawicz CM, Zisman TL. The microbiome and inflammatory bowel disease: is there a therapeutic role for fecal microbiota transplantation? Am J Gastroenterol. 2012 Oct;107(10):1452-9. doi: 10.1038/ajg.2012.93. PMID 23034604
- [Derived] Damman CJ, Brittnacher MJ, Westerhoff M, Hayden HS, Radey M, Hager KR, Marquis SR, Miller SI, Zisman TL. Low Level Engraftment and Improvement following a Single Colonoscopic Administration of Fecal Microbiota to Patients with Ulcerative Colitis. PLoS One. 2015 Aug 19;10(8):e0133925. doi: 10.1371/journal.pone.0133925. eCollection 2015. PMID 26288277